CLINICAL TRIAL: NCT00887055
Title: Bi-ventricular Capture Verification Study
Brief Title: OPTIMA Bi-ventricular Capture Verification Study
Status: Withdrawn | Type: Observational
Why Stopped: never started
Sponsor: Guidant Corporation (Industry)
Other Study IDs: OPTIMA
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: CRT device

SUMMARY:
The purpose of this study is to characterize the morphology (shape) of the intracardiac electrograms(EGM) from patients with a resynchronization therapy device.

DETAILED DESCRIPTION:
morphology of EGM during loss of capture in either right ventricle (RV) or left ventricle (LV) at different AV delays and LV offsets and during exercise. These EGM signals will be used to design and develop improved automatic threshold and automatic capture algorithms for CRT defibrillators (CRT-D). As well, the data collected from the study will be used to to develop other automatic algorithms for CRT-D, such as pacing parameter optimization.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent indicating a willingness to participate, have indications for and have been implanted with a Guidant Renewal 4 CRT-D device

Exclusion Criteria:

* Patients in atrial fibrillation that cannot be cardioverted for the study, sustained uncontrolled ventricular tachycardia (VT), sinus rhythm < 40 bpm or > 100 bpm, complete AV node block, AV node ablation, Severe aortic valve stenosis (valve area < 1.0 cm squared), frequent ectopic beats that would preclude adequate testing, lead in the great cardiac vein, women who are pregnant or who plan to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francois Philippon, MD, Principal Investigator — Hopital Laval, 2725 Chemin Ste-Foy, Ste-Foy, Quebec, Canada G1V 4G5 418-656-8711
Locations (1):
- Hopital Laval, Ste-Foy, Quebec, Canada